CLINICAL TRIAL: NCT03006848
Title: A Phase II Trial of Avelumab, A Fully Human Antibody That Targets Cells Expressing PD-L1, in Patients With Recurrent or Progressive Osteosarcoma
Brief Title: A Phase II Trial of Avelumab in Patients With Recurrent or Progressive Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Pfizer (Industry); Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSTPDL1; Pfizer W1211733 (OSTPDL1) (Other Grant/Funding Number: Pfizer, Inc.); Gateway RESAG (Other Grant/Funding Number: Gateway for Cancer Research)
Record Dates: First submitted 2016-12-22; First posted 2016-12-30 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Osteosarcoma
Keywords: Osteosarcoma; PD-L1; Immunotherapy
MeSH Terms: conditions — Osteosarcoma | interventions — avelumab; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab (Experimental): All participants with recurrent/refractory osteosarcoma who consent to the study.
  Interventions: Avelumab and quality of life questionnaires.
  Interventions: Drug: Avelumab; Other: Questionnaires

INTERVENTIONS:
Drug: Avelumab — Patients will be administered avelumab at a dose of 10 mg/kg intravenously (IV) over 60 minutes on days 1 and 15 of each cycle, with a cycle lasting 28 days. Patients will receive avelumab every 2 weeks in cycles of 28 days for up to 24 months, or 26 cycles.
  Other Names: MSB0010718C; anti-PD-L1
Other: Questionnaires — To assess quality of life, patients will complete questionnaires at four time points.
  Other Names: PROMIS Pediatric Profile; PROMIS Adult Profile

SUMMARY:
This clinical trial seeks to determine if avelumab will be effective in facilitating removal of all gross tumor in the event of a relapse of osteosarcoma in pediatric patients. Avelumab will be evaluated using dosing that has previously been determined in adult studies.

Primary Objectives:

* To estimate the response rate to 4 cycles of avelumab in patients with recurrent or progressive osteosarcoma.
* To estimate the 16-week progression free survival of patients with recurrent or progressive osteosarcoma after treatment with avelumab.

Secondary Objective:

* To describe the toxicities associated with the administration of avelumab in patients with recurrent or progressive osteosarcoma.
* To assess the quality of life of patients with recurrent or progressive osteosarcoma undergoing treatment with avelumab, and to explore relationships between clinical factors and patient-reported health-related quality of life (HRQOL) outcomes.

Exploratory Objectives:

* To explore factors associated with response in patients treated with avelumab after recurrent or progressive osteosarcoma (e.g. tumor PD-L1 expression).
* To measure parameters of immune activation including subsets of peripheral blood mononuclear cells (PBMCs) and serum markers of immune activation.
* To evaluate the role of T-cells in immune checkpoint blockade via measures of cell proliferation, co-inhibitory receptor expression on CD8 T cells, T cell repertoire, and epigenetic programming.

DETAILED DESCRIPTION:
This is a Phase 2 study using a traditional Simon two-stage design. Patients 12 years or greater with recurrent/refractory osteosarcoma will be administered avelumab at a dose of 10 mg/kg intravenously (IV) over 60 minutes on days 1 and 15 of each cycle, with a cycle lasting 28 days.

Patients will receive avelumab every 2 weeks in cycles of 28 days for up to 24 months, or 26 cycles. Progression free survival and response to therapy after 4 cycles of treatment will be assessed. In addition, the toxicity profile of avelumab in this population will be closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > 12 years of age but < 50 years of age at the time of enrollment.
* Patients must have histologic verification of osteosarcoma at initial diagnosis or relapse.
* Patients must have had evidence of having relapsed, progressed or become refractory to conventional therapy.
* Patients must have measurable disease, documented by clinical, radiographic or histologic criteria. Disease must be bi-dimensionally measurable by computed tomography (CT) or magnetic resonance imaging (MRI).
* Patients must have a performance status of ≥ 50 using the Karnofsky scale for patients > 16 years of age and the Lansky scale for patients ≤ 16 years of age.
* Patients must have a life expectancy of ≥ 6 weeks.
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

  1. Myelosuppressive chemotherapy: must not have received within 3 weeks of entry onto this study.
  2. Biologic (anti-neoplastic agent): at least 7 days since the completion of therapy with a biologic agent.
  3. Immunotherapies: at least 42 days must have elapsed since a prior therapy that included a monoclonal antibody or any other type of immunotherapy (e.g. chimeric antigen receptor (CAR) T cell therapy).
  4. Radiation therapy (RT): ≥ 2 weeks for local palliative RT (small port); ≥ 6 months must have elapsed if prior craniospinal RT or if ≥ 50% radiation of the pelvis; ≥ 6 weeks must have elapsed if other substantial bone marrow (BM) radiation.
* Organ Function Requirements:

  1. Adequate bone marrow function defined as:

     * Peripheral absolute neutrophil count (ANC) ≥ 1500/mm3
     * Platelet count ≥ 100,000/mm3 (transfusion independent)
     * Hemoglobin ≥ 9.0 g/dL (may receive RBC transfusions)
  2. Adequate renal function defined as:

     * Creatinine clearance or radioisotope GFR ≥70 mL/min/1.73m2 OR
     * Serum creatinine based on age/gender as follows: (threshold creatinine values were derived from the Schwartz formula for estimating GFR).

       * Age is: 12 to <13 years, then maximum creatinine is 1.2 mg/DL for male and female.
       * Age is: 13 to <16 years, then maximum creatinine is 1.5 mg/DL for male and 1.4 mg/DL for female.
       * Age is: ≥16 years, then maximum creatinine is 1.7 mg/DL for male and 1.4 mg/DL for female.
  3. Adequate liver function defined as:

     * Total Bilirubin ≤ 1.5x the institutional upper limit of normal (IULN) for age
     * ALT (SGPT) and AST (SGOT) < 2.5 x IULN for age (or < 5 x IULN for patients with documented metastatic disease to the liver)
     * Serum albumin > 2 g/dL
  4. Serum lipase ≤ upper limit of normal (IULN).
  5. Patients must have documented pulse oximetry ≥ 92% on room air.
* Female patients of childbearing potential must have a negative serum or urine pregnancy test within 7 days of enrollment.
* Male or female patients who are sexually active and of reproductive potential must agree to use an effective contraceptive method throughout the study and for at least 60 days after last avelumab treatment administration. Abstinence is an acceptable form of contraception.
* Patients must not currently be using other investigational agents.
* Patients must not currently be using other anti-cancer agent.
* Patients must be able to comply with the safety monitoring of the study in the opinion of the investigator.
* Written, informed consent and assent following Institutional Review Board, NCI, FDA and OHRP guidelines.

Exclusion Criteria:

* Central nervous system (CNS) metastases.
* Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* Active infection requiring systemic therapy.
* Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive).
* Patient who has received vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3).
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II, see Appendix II), or serious cardiac arrhythmia requiring medication.
* Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable
* Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Patients with active diarrhea > CTCAE v4.03 Grade 2.
* Patients who have previously received a prior organ transplantation, including allogeneic stem cell transplantation.
* Female patients who are pregnant or actively breastfeeding.
* Patients who have previously received anti-PD1 or anti-PD-L1 therapy. Patients who have previously received anti-CTLA-4 therapy (e.g. ipilimumab) are eligible for study.

Ages: 12 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Bishop, MD, MS, Principal Investigator — St. Jude Children's Research Hospital
Locations (4):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 19 patients were enrolled on the study from February 2017 to April 2021
Pre-assignment Details: 18 out of 19 enrolled patients received treatment. The patient who did not receive treatment was found to be ineligible and thus was a screen failure.
Groups:
- Avelumab: All participants with recurrent/refractory osteosarcoma who consent to the study.
  Interventions: Avelumab and quality of life questionnaires.
  Avelumab: Patients will be administered avelumab at a dose of 10 mg/kg intravenously (IV) over 60 minutes on days 1 and 15 of each cycle, with a cycle lasting 28 days. Patients will receive avelumab every 2 weeks in cycles of 28 days for up to 24 months, or 26 cycles.
  Questionnaires: To assess quality of life, patients will complete questionnaires at four time points.
Period: Overall Study
Arm/Group | Avelumab
Started | 18
Completed | 0
Not Completed | 18
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 16

BASELINE CHARACTERISTICS:
Units Other Than Participants: years
Arm/Group | Avelumab
Number analyzed (Participants) | 18
Number analyzed (years) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.0 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 14
  Race: Black | 2
  Race: Declined Respond | 1
  Race: Unknown | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States: St. Jude Children's Research Hospital | 14
  United States: Memorial Sloan-Kettering Cancer Center | 2
  United States: Children's Hospital of Los Angeles | 1
  United States: Texas Children's Research Hospital | 1
Disease Status at time of enrollment [Count of Participants; unit: Participants]
  Progressive Disease | 13
  Recurrent Disease | 5

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: The study is designed by treating RECIST response [complete response + partial response (CR+PR)] after 4-cycle treatment of avelumab and the 16-week progression-free survival (PFS) as dual binary endpoints. Patients who fail to be evaluated at the end of the 4-cycle will be counted as failure.
Time Frame: At the end of 4 cycles of avelumab (approximately 4 months)
Population: RECIST response [complete response + partial response (CR+PR)]
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab
Number analyzed (Participants) | 18
percentage of participants | 0 [0 to 0]

2. Primary Outcome: Progression-free Survival
Description: as for outcome 1
Time Frame: At the end of 4 cycles of avelumab (approximately 4 months)
Population: Of the 18 eligible patients who received treatment, 17 patients had disease progression while on study and one patient died off study.
Measure: Median (95% Confidence Interval); unit: percentage of weeks
Groups:
- Progression-free Survival: The study is designed by treating RECIST response [complete response + partial response (CR+PR)] after 4-cycle treatment of avelumab and the 16-week progression-free survival (PFS) as dual binary endpoints. Patients who fail to be evaluated at the end of the 4-cycle will be counted as failure.
Arm/Group | Progression-free Survival
Number analyzed (Participants) | 18
percentage of weeks | 8.0 [6.7 to 9.1]

3. Secondary Outcome: Target Toxicities
Description: Target toxicities for avelumab treatment are defined as any grade 3-5 dyspnea, infusion-related reactions, or immune related adverse events at least possibly attributable to the agent observed anytime during the 26-cycle treatment period that a patient is on study (including the period between off treatment and off study).
Time Frame: At the end of treatment (up to 2 years after enrollment of last participant)
Population: [Not Specified]
Measure: Number; unit: participants
Groups:
- Target Toxicities: Target toxicities for avelumab treatment are defined as any grade 3-5 dyspnea, infusion-related reactions, or immune related adverse events at least possibly attributable to the agent observed anytime during the 26-cycle treatment period that a patient is on study (including the period between off treatment and off study).
Arm/Group | Target Toxicities
Number analyzed (Participants) | 18
participants
  Dyspnea | 2
  Infection and infestations | 1
  Metabolism and nutrition disorders | 2
  Blood and lymphatic system disorders | 1
  Cardiac disorders | 1
  Investigations | 2

4. Other Pre Specified Outcome: Factors Associated With Response
Description: Logistic regression analysis will be conducted to explore factors which may associate with response.
Time Frame: Following completion of therapy for last participant (up to 2 years after enrollment)
Population: [Not Specified]
Groups:
- Factors Associated With Response: Logistic regression analysis will be conducted to explore factors which may associate with response.
Arm/Group | Factors Associated With Response
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Change in Parameters of Immune Activation
Description: Descriptive statistics will be provided.
Time Frame: Baseline prior to start of therapy and following 2 cycles of therapy (up to 8 weeks after last enrollment)
Population: [Not Specified]
Groups:
- Change in Parameters of Immune Activation: Descriptive statistics will be provided.
Arm/Group | Change in Parameters of Immune Activation
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Change in Cell Proliferation
Description: Descriptive statistics will be provided.
Time Frame: Baseline prior to start of therapy and after completion of therapy (approximately 2 years after last participant enrollment).
Population: [Not Specified]
Groups:
- Change in Cell Proliferation: Descriptive statistics will be provided.
Arm/Group | Change in Cell Proliferation
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Change in Co-inhibitory Receptor Expression on CD8 T Cells
Description: Descriptive statistics will be provided.
Time Frame: as for outcome 6
Population: [Not Specified]
Groups:
- Change in Co-inhibitory Receptor Expression on CD8 T Cells: Descriptive statistics will be provided.
Arm/Group | Change in Co-inhibitory Receptor Expression on CD8 T Cells
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Change in Quality of Life
Description: Participants will self-report their quality of life through PROMIS questionnaires, either the Pediatric Profile (ages 8 to 17 years) or the Adult Profile (age 18 years or older). The change in age-normed T-scores will be reported. Mixed effect models will be performed to assess changes in quality of life over time.
Time Frame: From baseline prior to start of treatment through the end of avelumab therapy (up to approximately 2 years)
Population: [Not Specified]
Groups:
- Change in Quality of Life: Participants will self-report their quality of life through PROMIS questionnaires, either the Pediatric Profile (ages 8 to 17 years) or the Adult Profile (age 18 years or older). The change in age-normed T-scores will be reported. Mixed effect models will be performed to assess changes in quality of life over time.
Arm/Group | Change in Quality of Life
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Acute adverse events were collected from study enrollment up to 4 weeks after completion of chemotherapy/radiation therapy, whichever came last. Long term toxicity was captured at every visit up to 3 years from study enrollment.
Description: [Not specified]
Groups:
- Avelumab: [Not specified]
Arm/Group | Avelumab
All-Cause Mortality (participants affected / at risk) | 3/18
Serious Adverse Events (participants affected / at risk) | 7/18
Other Adverse Events (participants affected / at risk) | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab (N=18)
Blood and lymphatic system disorders (Vascular disorders) | 1 (1) — Thromboembolic event
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Neoplasms benign, malignant and unspecified
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Dyspnea
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Bronchopulmonary hemorrhage
Infections and infestations (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Lung infection
Nervous system disorders (Nervous system disorders) | 1 (1) — Stroke
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) — Abdominal pain
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) — Hyponatremia
Investigations (Investigations) | 1 (1) — Aspartate aminotransferase increased
Investigations (Investigations) | 1 (1) — Alanine aminotransferase increased
Cardiac disorders (Cardiac disorders) | 1 (1) — Pericardial effusion
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab (N=18)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) — Anemia
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (2) — Blood and lymphatic system disorders - Other
Cardiac disorders (Cardiac disorders) | 1 (1) — Sinus tachycardia
Cardiac disorders (Cardiac disorders) | 1 (1) — Pericardial tamponade
Endocrine disorders (Endocrine disorders) | 1 (2) — Hyperthyroidism
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) — Diarrhea
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) — Gastritis
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3) — Constipation
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3) — Nausea
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (2) — Abdominal pain
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) — Hemorrhoids
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) — Rectal pain
General disorders and administration site conditions (General disorders) | 1 (2) — Fever
General disorders and administration site conditions (General disorders) | 3 (7) — Pain
General disorders and administration site conditions (General disorders) | 1 (1) — Fatigue
General disorders and administration site conditions (General disorders) | 1 (2) — Non-cardiac chest pain
General disorders and administration site conditions (General disorders) | 1 (1) — Gait disturbance
Immune system disorders (Immune system disorders) | 1 (1) — Autoimmune disorder
Infections and infestations (Infections and infestations) | 2 (2) — Lung infection
Infections and infestations (Infections and infestations) | 1 (1) — Urinary tract infection
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2) — Fall
Investigations (Investigations) | 2 (2) — Alkaline phosphatase increased
Investigations (Investigations) | 1 (1) — Aspartate aminotransferase increased
Investigations (Investigations) | 2 (3) — Alanine aminotransferase increased
Investigations (Investigations) | 1 (1) — Blood bilirubin increased
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) — Hyperglycemia
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (2) — Hypokalemia
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) — Hyponatremia
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 (4) — Back pain
Nervous system disorders (Nervous system disorders) | 1 (1) — Paresthesia
Nervous system disorders (Nervous system disorders) | 1 (3) — Peripheral sensory neuropathy
Nervous system disorders (Nervous system disorders) | 1 (2) — Headache
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) — Proteinuria
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dyspnea
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pleuritic pain
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Allergic rhinitis
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumonitis
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Bronchopulmonary hemorrhage
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Cough
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) — Rash acneiform
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (2) — Alopecia

LIMITATIONS AND CAVEATS:
One patient changed administration schedule for C2D15 in cycle 2 due to family vacation plan. The variance in dates was submitted to IRB and the patient was approved to continue on treatment when returns from the trip.

One patient was unable to travel from Puerto Rico due to hurricane devastation. Dose C2D15 skipped in cycle 2.

Medications were given one or two day(s) earlier or later than the scheduled date for a few patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT03006848/Prot_SAP_000.pdf